CLINICAL TRIAL: NCT05945121
Title: Cardio-Oncology Prehabilitation Program to Improve Cardiac Reserve in High-Risk Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Prehabilitation Program to Improve Cardiac Reserve in High-Risk Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.004; HUM00223835 (Other: University of Michigan); U24HL157560 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-07-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardio-oncology program (Experimental): The cardio-oncology program consists of a multimodal approach, which includes individualized exercise prescription following a detailed CV assessment and medical management of CV risk factors occurring over 8 weeks.
  Interventions: Other: Cardio-oncology program

INTERVENTIONS:
Other: Cardio-oncology program — Consented patients will undergo an initial CV evaluation as part of standard of care then participate in an 8-week at-home, personalized exercise intervention followed by an additional CV assessment prior to HSCT (after 8-weeks)

SUMMARY:
To assess the feasibility and preliminary effectiveness of a Cardio-Oncology Prehabilitation program in patients at high-risk of developing Cardiovascular (CV) events in improving Cardiorespiratory fitness (CRF) and reducing acute CV complications in Hematopoietic stem cell transplant (HSCT) recipients.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older
* Referred for HSCT evaluation
* Presence of least one CV risk factor at enrollment (hypertension, hyperlipidemia, atrial fibrillation, obesity, heart failure, history of coronary artery disease, diabetes)
* Able to ambulate unassisted
* Ability to understand and the willingness to sign a written informed consent
* Ability to use Polar Flow heart rate application

Exclusion Criteria:

* Severe anemia (hemoglobin <7 gm/dl)
* Untreated high-risk coronary artery disease (left main, triple vessel disease)
* Severe aortic stenosis
* Recent fracture as assessed via self-report
* Gross balance deficits
* Severe pain with basic movement
* Unable to ambulate unassisted or exercise
* NYHA class IV heart failure
* Adults unable to give consent, pregnant women, and prisoners are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (Recruitment Rate). | 8 weeks post enrollment
  Percent of eligible participants who are screened and give informed consent
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (retention Rates). | 8 weeks post enrollment
  percentage of enrolled participants who complete pre-post CV assessments
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (Duration of Recruitment). | 8 weeks post enrollment
  the number of participants recruited per month
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (time to implement study protocol). | 8 weeks post enrollment
  the average amount of time required for participants to complete initial and follow-up CV assessments
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (adherence to program- Days). | 8 weeks post enrollment
  The percentage of days of exercised out of 24 days recommended over the 8 weeks for both aerobic and resistance activities.
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (adherence to program- Time). | 8 weeks post enrollment
  The average duration (min) of aerobic and resistance workouts over the course of the intervention.
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (adherence to program- Missing data). | 8 weeks post enrollment
  the percentage of missing data from study questionnaires.
Feasibility of a cardio-oncology prehabilitation program in high-risk HSCT candidates (overall satisfaction). | 8 weeks post enrollment
  Assessed qualitatively with in-depth, semi-structured, one-to-one exit interviews with participants. A member of the research team experienced with telephone interviews, but not involved in intervention delivery, will contact all patients within 1 week after completion of the final follow-up assessment.The researcher will facilitate the interviews using a conversational-style approach whilst referring to a topic guide. Topics will focus on patients' perceived expectations, benefits, motives, and barriers to the program. The researcher will additionally ask questions regarding reasons for non-adherence to the exercise intervention, and reasons for dropout amongst discontinuing patients. The topic guide will be used flexibly to allow patients to raise additional issues which they consider important to the study. Interviews will be recorded with participants knowledge and then transcribed, coded, and assessed for relevant themes and recommendations using iterative thematic analysis
Preliminary effectiveness of an 8-week cardio-oncology prehabilitation on measures of CRF in high-risk HSCT candidates (change in anaerobic threshold). | 8 weeks post enrollment
  change in anaerobic threshold from pre to post intervention reported in L/min
Preliminary effectiveness of an 8-week cardio-oncology prehabilitation on measures of CRF in high-risk HSCT candidates (change in VO2peak). | 8 weeks post enrollment
  change in VO2peak from pre to post intervention reported in ml/kg/min
Preliminary effectiveness of an 8-week cardio-oncology prehabilitation on measures of CRF in high-risk HSCT candidates (comparison of V02 peak to predicted). | 8 weeks post enrollment
  Comparison of V02 peak assessed after intervention in comparison to the predicted values reported as the percent difference between the values
Preliminary effectiveness of an 8-week cardio-oncology prehabilitation on measures of CRF in high-risk HSCT candidates (RER). | 8 weeks post enrollment
  change in RER (a ratio between cardiac dioxide output (VCO2)/oxygen uptake (VO2)) from pre to post intervention reported as the percent difference between the values
Preliminary effectiveness of an 8-week cardio-oncology prehabilitation on measures of CRF in high-risk HSCT candidates (VE/VC02 slope). | 8 weeks post enrollment
  Change in VE/VC02 slope (defined as the change in minute ventilation per unit of carbon dioxide production) from pre to post intervention

SECONDARY OUTCOMES:
Symptom assessment scores after an 8-week cardio-oncology prehabilitation program. | 8 weeks post enrollment
  Frequency and severity of cardiovascular symptoms (fatigue, shortness of breath, edema) will be assessed using the short Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health. Items are grouped into the four domains; Physical limitation, Symptom frequency, Quality of life, and Social limitation.
Changes in patient reported quality of life after an 8-week cardio-oncology prehabilitation program | 8 weeks post enrollment
  Overall quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Responses are given on a single-item ranging in score from 0 to 100. A high scale score represents a higher response level.
Difference in biomarkers after an 8-week cardio-oncology prehabilitation program | 8 weeks post enrollment
  High-sensitivity troponin-I (RayBiotech), B-type natriuretic peptide (BNP) (RayBiotech), and soluble urokinase plasminogen activator receptor (suPAR) (Virogates) will be measured in residual serum samples collected as part of usual care using enzyme-linked immunosorbent assays.
Change in patient HSCT eligibility after an 8-week cardio-oncology prehabilitation program | 8 weeks post enrollment
  We will calculate the percentage of participants evaluated who end up being eligible for HSCT and compare rates to the number of participants who are referred to cardio-oncology, do not receive the intervention, and are considered ineligible.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No